CLINICAL TRIAL: NCT04761107
Title: Mitigating Risk of COVID-19 for Clinical Management of Genitourinary Diseases
Brief Title: Impact of COVID-19 on GU Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ashutosh Kumar Tewari, Professor and System Chair, Urology, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 20-1053; STUDY-20-01467 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Infection; Genitourinary Cancer; Benign Urologic Conditions
Keywords: COVID-19 Infection; Biomarkers; Prostate cancer, BPH; Bladder cancer, Urinary tract infection; Kidney stone, Kidney cancer; Malignant disease
MeSH Terms: conditions — COVID-19; Urogenital Neoplasms; Prostatic Neoplasms; Prostatic Hyperplasia; Urinary Bladder Neoplasms; Urinary Tract Infections; Kidney Calculi; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Peripheral blood - plasma and serum for PBMCs and aliquots.
  2. Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GU participants with active or past infection of SARS-Co-V-2: GU patients from medical records with active or past infection of SARS-Co-V-2

SUMMARY:
The purpose of this research study is to identify patients with GU disease with active or past COVID-19 infection.

Participants will be asked to:

* Complete an Online COVID-19 Questionnaire.
* Disclose if the patient has or had Genitourinary cancer or benign urologic condition
* Provide urine specimen for research
* Provide 4 tablespoons of blood for testing blood for research.
* Provide permission to access medical records, such as patient lab results, medical history, imaging reports, etc.

DETAILED DESCRIPTION:
COVID-19 has a higher incidence in males compared to females and cancer patients have a higher risk of contracting COVID-19, and developing complications, and deteriorate more rapidly. COVID19 pandemic poses significant challenges in clinical decision-making, which has impacted management of GU patients. In order to mitigate the risk associated with COVID19 pandemic while also providing the best clinical care for patients a screening approach is essential. Clinicians taking care of cancer patients will be expected not only to understand impact of COVID19 but also incorporate a triage tool to decide which patients need immediate treatment. This prospective study presented in this IRB is about establishing a screening tool for GU patients with pre-existing cancer or with benign urological disease (e.g. BPH, kidney stone, bladder infection, urinary tract infections etc) and for those who are dealing with decisions for biopsy, active surveillance, surgery, radiation, hormonal and chemotherapy.

The study team is expecting to enroll 15240 subjects under this study.

Procedures involved in the study:

1. Consenting patients for the study.
2. Screening/Baseline REDCap survey to determine their COVID-19 symptoms.
3. Blood sample collection: This will be obtained for research studies including immune monitoring assays
4. Urine sample collection for bio-marker analysis.
5. Data collection from medical records, such as:

   * Clinical diagnoses, including date of confirmation of SARS-CoV-2 infection
   * Any pertinent medical history, including concomitant medications, and comorbidities that pre- date enrollment in the study, or that occur during enrollment in the study
   * Laboratory values from time of blood procurement
   * All imaging (X-ray, MRI, CAT, PAT, PSMA, Ultrasound, and Pathology etc.) performed from time of initial diagnosis until death, and any needed imaging that pre- date enrollment that may serve as a comparative to pre/post treatment imaging.
   * Collection time of samples in relation to study treatment
   * Demographic data
   * REDCap questionnaire, COVID-19 symptoms and severity of the symptoms

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be men and women 40 years of age or older
* Subjects at risk or with GU cancer (Prostate, Bladder, Kidney)
* Subjects with benign GU disorders ( BPH, UTI, Bladder infection and kidney stone)
* Subjects must have a GU disease that requires clinic visit as determined by physician or healthcare provider following a telehealth appointment
* Willing and able to provide blood and urine samples
* Willing and able to complete a questionnaire to determine the COVID-19 symptoms.
* Willing and able to sign informed consent form

Exclusion Criteria:

* Men and women below 40 years of age
* Subjects do not have a GU disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the Urology Department at Mount Sinai.
Sampling Method: Probability Sample
Enrollment: 15240 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a new diagnosis of GU | Day 1
  Proportion of patients with a new diagnosis of GU cancer and with active or past infection with SARS-Co-V-2

SECONDARY OUTCOMES:
Proportion of GU cancer patients, with active disease or in remission | Day 1
  Proportion of GU cancer patients, with active disease or in remission and with active or past infection with SARS-Co-V-2
Proportion of patients with the benign urologic condition | Day 1
  Proportion of patients with the benign urologic condition and with active or past infection with SARS-Co-V-2

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh K Tewari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Dimple Chakravarty, PhD, Study Director — Icahn School of Medicine at Mount Sinai; Sujit S Nair, PhD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Chakravarty D, Nair SS, Hammouda N, Ratnani P, Gharib Y, Wagaskar V, Mohamed N, Lundon D, Dovey Z, Kyprianou N, Tewari AK. Sex differences in SARS-CoV-2 infection rates and the potential link to prostate cancer. Commun Biol. 2020 Jul 8;3(1):374. doi: 10.1038/s42003-020-1088-9. PMID 32641750
- [Background] Lundon DJ, Kelly BD, Nair S, Bolton DM, Kyprianou N, Wiklund P, Tewari A. Early mortality risk stratification after SARS-CoV-2 infection. Med Intensiva (Engl Ed). 2020 Jul 4;45(8):e40-2. doi: 10.1016/j.medin.2020.06.011. Online ahead of print. No abstract available. PMID 32912654
- [Background] Pavlova IP, Nair SS, Kyprianou N, Tewari AK. The Rapid Coronavirus Antibody Test: Can We Improve Accuracy? Front Med (Lausanne). 2020 Sep 2;7:569. doi: 10.3389/fmed.2020.00569. eCollection 2020. No abstract available. PMID 32984390
- [Background] Theise ND, Arment AR, Chakravarty D, Gregg JMH, Jacobson IM, Jung KH, Nair SS, Tewari AK, Thurston AW, Van Drie J, Westover JB. Clinical stage molecule PT150 is a modulator of glucocorticoid and androgen receptors with antiviral activity against SARS-CoV-2. Cell Cycle. 2020 Dec;19(24):3632-3638. doi: 10.1080/15384101.2020.1859752. Epub 2020 Dec 11. PMID 33305659